CLINICAL TRIAL: NCT04041297
Title: Evaluation of Non-Small Cell Lung Cancer Patients' Oxygen Uptake On-kinetics at Cycle-ergometer During Prehabilitation
Brief Title: Evaluation of NSCLC Patients' Oxygen Uptake On-kinetics at Cycle-ergometer During Prehabilitation
Acronym: Preo-Kinetics
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: Preo-Kinetics
Record Dates: First submitted 2019-07-28; First posted 2019-08-01 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Preoperative training; Prehabilitation; oxygen-uptake kinetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Preoperative Pulmonary Rehabilitation — Each prehabilitation session will last approximately 90 minutes and will include:
  Endurance training at the ventilatory threshold, determined according to the initial CPET. The first session will last for 15 to 20 minutes then increase by 5 minutes each session to reach 45 minutes in total (including a 5-minute warm-up and 5 minutes of active recovery). The intensity will then increase by 5 or 10 W, as could be tolerated;
  Peripheral muscle strengthening at 60% to 70% of the 1-repetition maximum of 3 main components (quadriceps press, whole-leg extension, and upper limb pull down). Three sets of 12 movements will carry out for each exercise and the load will increase weekly as tolerated;
  Inspiratory muscle training using a threshold calibrated to at least 30% of the MIP. Patients will be encouraged to carry out 15 minutes of independent training daily and to increase the resistance regularly.
  Education to bronchial drainage techniques as well as directed coughing.

SUMMARY:
In developed countries cancer has become the second leading cause of death after cardiovascular disease. The lung is a particularly exposed organ since broncho-pulmonary cancers rank second in terms of incidence, and the first rank in terms of mortality of all cancers listed in like reported in United States.

Lung resection surgery is currently the recommended curative treatment for the early stages of non-small cell lung cancer (NSCLC). Despite this preferred indication, some patients can not be eligible for surgery because of their cardiovascular or respiratory comorbidities or their impaired functional capacity.

Thus, the evaluation of aerobic capacity through cardiopulmonary exercise testing (CPET) of patients estimated at risk of postoperative complication is now recommended to estimate the level of predictive risk associated. The American Thoracic Society and the European Respiratory Socitety agree on thresholds of <10 and> 20 ml/kg/min of maximum oxygen uptake (VO2peak) respectively determining a high or low postoperative risk, between these two thresholds risk is considered moderate.

Aerobic capacity is traditionally expressed in terms of maximum oxygen uptake (VO2max or VO2peak) evaluated during an incremental CPET. In patients with significant respiratory impairment, these tests are often limited by ventilation and sub-maximally on the metabolic or cardiac parameters. However, the analysis of the VO2 kinetic during a constant-intensity test of moderate intensity is also a relevant way of measuring aerobic conditioning. Indeed, the time constant (τ) of phase II of VO2 kinetics (VO2τ) is a marker that closely reflects the adjustment of oxidative metabolism in skeletal muscle. Analysis of the kinetic parameters of the cardio-respiratory response to exercise has been shown to be reproducible and training-sensitive in patients with chronic obstructive pulmonary disease (COPD). The value of VO2τ was also reported to be strongly correlated with markers of severity and prognosis in COPD patients. Previous work has shown that exercise training can improve the speed of the VO2 kinetic response in COPD patients as well as in healthy subjects.

To date, no study to our knowledge has evaluated the kinetics of the cardiorespiratory response during moderate intensity constant-load test in patients with NSCLC. In this context, this work aims to evaluate the applicability of this measure as well as its evolution during a preoperative exercise training program in patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old;
* Beneficiary of a social security scheme;
* Non-Small Cell Lung Cancer or suspicion of bronchial neoplasia;
* Addressed to respiratory rehabilitation in a preoperative setting with a moderate to high risk estimate (VO2peak < 20 ml/kg/min);
* Intervention date not established when included in the program or ≥ 5 wk.

Exclusion Criteria:

* Patient under guardianship;
* Pregnant or lactating woman;
* Cardiological contraindication to training;
* Neoadjuvant radio-chemotherapy;
* Refusal to carry out a training program in a rehabilitation center;
* Orthopedic, neurological, vascular or neuromuscular pathology limiting training;
* Exacerbation or deterioration of the general condition requiring stopping the preoperative re-training program;
* Modification of the therapeutic project at a multidisciplinary consultation meeting requiring the cessation of rehabilitation or participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred in the ADIR Association for a preoperative pulmonary rehabilitation program in preparation for lung resection surgery for non-small cell lung cancer are concerned.
  They are contacted by one of the rehabilitation physiotherapists to carry out an inclusion consultation in the respiratory rehabilitation program. During this session, the study is presented to them and their consent to study is collected.
  Participation in or refusal of the study does not affect the overall standard of care provided during the program.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Phase II time constant of Oxygen uptake kinetics (VO2τ), during a constant load test on a cyclo ergometer | before the preoperative training program
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). VO2 uptake is collected cycle by cycle by a gas exchange analysis system (Vyntus® CPX, CareFusion, Hoechberg, Germany)
Phase II time constant of Oxygen uptake kinetics (VO2τ), during a constant load test on a cyclo ergometer | through preoperative training program completion (15 sessions), an average of 1 month
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). VO2 uptake is collected cycle by cycle by a gas exchange analysis system (Vyntus® CPX, CareFusion, Hoechberg, Germany)

SECONDARY OUTCOMES:
Phase II time constant of heart rate kinetics (HRτ), during a constant load test on a cyclo ergometer | before the preoperative training program
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). Heart rate is continuously collected by a 12-lead electrocardiogram dyspositif (EC Sense Lexor, Cardiolex, Solna, Sweden)
Phase II time constant of heart rate kinetics (HRτ), during a constant load test on a cyclo ergometer | through preoperative training program completion (15 sessions), an average of 1 month
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). Heart rate is continuously collected by a 12-lead electrocardiogram dyspositif (EC Sense Lexor, Cardiolex, Solna, Sweden)
Steady state oxygen uptake (VO2ss), during a constant load test on a cyclo ergometer | before the preoperative training program
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). VO2 uptake is collected cycle by cycle by a gas exchange analysis system (Vyntus® CPX, CareFusion, Hoechberg, Germany)
Steady state oxygen uptake (VO2ss), during a constant load test on a cyclo ergometer | through preoperative training program completion (15 sessions), an average of 1 month
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). VO2 uptake is collected cycle by cycle by a gas exchange analysis system (Vyntus® CPX, CareFusion, Hoechberg, Germany)
Steady-state heart rate (HRss), during a constant load test on a cyclo ergometer | before the preoperative training program
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). Heart rate is continuously collected by a 12-lead electrocardiogram dyspositif (EC Sense Lexor, Cardiolex, Solna, Sweden)
Steady-state heart rate (HRss), during a constant load test on a cyclo ergometer | through preoperative training program completion (15 sessions), an average of 1 month
  maintaining a constant power corresponding to 80% of the anaerobic threshold or failing that 50% of the VO2peak obtained at the incremental CPET (Puente-Maestu et al. 2001). Heart rate is continuously collected by a 12-lead electrocardiogram dyspositif (EC Sense Lexor, Cardiolex, Solna, Sweden)
Peak oxygen uptake (VO2peak) obtained during the incremental cardiopulmonary exercise testing | before the preoperative training program
  Incremental cardiopulmonary exercise testing (CPET) standardized on the statement of the American Thoracic Society and American College of Chest Physicians 2003, on cyclo-ergometer. Performed during the evaluation process before pulmonary resection surgery and allows to refer patients at risk to preoperative retraining.
Peak oxygen uptake (VO2peak) obtained during the incremental cardiopulmonary exercise testing | through preoperative training program completion (15 sessions), an average of 1 month
  Incremental cardiopulmonary exercise testing (CPET) standardized on the statement of the American Thoracic Society and American College of Chest Physicians 2003, on cyclo-ergometer. Evaluation post preoperative exercise training to re-calculate postoperative risk.
Maximum heart rate (HRmax) reached during the incremental cardiopulmonary exercise testing | before the preoperative training program
  Incremental cardiopulmonary exercise testing (CPET) standardized on the statement of the American Thoracic Society and American College of Chest Physicians 2003, on cyclo-ergometer. Evaluation post preoperative exercise training to re-calculate postoperative risk.
Maximum heart rate (HRmax) reached during the incremental cardiopulmonary exercise testing | through preoperative training program completion (15 sessions), an average of 1 month
  Incremental cardiopulmonary exercise testing (CPET) standardized on the statement of the American Thoracic Society and American College of Chest Physicians 2003, on cyclo-ergometer. Evaluation post preoperative exercise training to re-calculate postoperative risk.

CONTACTS AND LOCATIONS:
Locations (1):
- ADIR Association, Bois-Guillaume, Normandy, France